CLINICAL TRIAL: NCT00040950
Title: A Multi-Center, Phase I, Open Label, Two Arm, Non-Randomized, Dose-Escalation, Study Of The Safety And Tolerability Of CPG 7909 In Patients Receiving Rituxan For Relapsed Or Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: Biological Therapy Plus Monoclonal Antibody Therapy in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069423; UCLA-0112032; CPGI-C004-CPG7909; NCI-G02-2086
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2003-07

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

INTERVENTIONS:
Biological: rituximab
Drug: agatolimod sodium

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Biological therapies such as CpG 7909 use different ways to stimulate the immune system and stop cancer cells from growing. Combining CpG 7909 with rituximab may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of CpG 7909 plus rituximab in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of subcutaneous and IV CpG 7909 when administered with rituximab in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the disease response in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of CpG 7909. Patients are sequentially assigned to 1 of 2 treatment groups.

* Group A: Patients receive rituximab IV over 4-5 hours followed by CpG 7909 IV over 2 hours on day 1. Courses repeat weekly for 4 weeks.
* Group B: Patients receive rituximab as above followed by CpG 7909 subcutaneously on day 1. Courses repeat weekly for 4 weeks.

Cohorts of 3-6 patients receive escalating doses of CpG 7909 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 6-48 patients (3-24 per treatment group) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD20+ B-cell non-Hodgkin's lymphoma (NHL)

  * CD20 positive by immunohistochemistry or flow cytometry
* Relapsed or refractory disease
* Bidimensionally measurable disease

  * Sole site of measurable disease within a previously irradiated field allowed provided there was disease progression at that site
* No pre-existing ascites or pleural effusions
* No known CNS involvement by NHL

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* Neutrophil count at least 1,000/mm3
* Platelet count at least 50,000/mm3

Hepatic:

* Bilirubin less than 2 mg/dL
* Transaminase less than 2 times upper limit of normal
* No hepatitis B or C

Renal:

* Creatinine less than 2 mg/dL

Cardiovascular:

* No significant cardiovascular disease
* No New York Heart Association class III congestive heart failure
* No myocardial infarction within the past 6 months
* No unstable angina
* No uncontrolled atrial or ventricular cardiac arrhythmias

Pulmonary:

* No concurrent significant pulmonary disease

Other:

* HIV negative
* No acute infection requiring antibiotics
* No fever over 38.2 degrees C within the past 3 days
* No other malignancy within the past 5 years except basal cell or noninvasive squamous cell skin cancer or carcinoma in situ of the cervix
* No pre-existing autoimmune disease or antibody-mediated disease, including:

  * Systemic lupus erythematosus
  * Rheumatoid arthritis
  * Multiple sclerosis
  * Sjogren's syndrome
  * Autoimmune thrombocytopenia
* Controlled thyroid disease allowed
* Concurrent autoantibodies without clinical autoimmune disease allowed
* No history of allergic reactions attributed to compounds of similar composition to study drugs
* No other medical history, including laboratory results, that would preclude study
* No suspected or confirmed poor compliance or mental instability that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior allogeneic transplantation
* More than 30 days since prior hematopoietic growth factors (e.g., filgrastim (G-CSF) or epoetin alfa)
* More than 30 days since prior immunotherapy
* More than 90 days since prior monoclonal antibodies as monotherapy for patients who were unresponsive to treatment (30 days for patients who responded to treatment and subsequently relapsed)
* No other concurrent biological agents
* No concurrent hematopoietic growth factors (e.g., G-CSF or epoetin alfa)

Chemotherapy:

* More than 30 days since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* More than 30 days since prior systemic corticosteroids
* No concurrent systemic corticosteroids

Radiotherapy:

* See Disease Characteristics
* More than 30 days since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* Recovered from prior therapy
* At least 6 months since prior coronary angioplasty
* More than 30 days since prior immunosuppressants
* More than 30 days since prior participation in an investigational drug study
* No concurrent immunosuppressants
* No concurrent anticoagulants except aspirin at doses no greater than 325 mg/day
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Leonard JP, Link BK, Emmanouilides C, Gregory SA, Weisdorf D, Andrey J, Hainsworth J, Sparano JA, Tsai DE, Horning S, Krieg AM, Weiner GJ. Phase I trial of toll-like receptor 9 agonist PF-3512676 with and following rituximab in patients with recurrent indolent and aggressive non Hodgkin's lymphoma. Clin Cancer Res. 2007 Oct 15;13(20):6168-74. doi: 10.1158/1078-0432.CCR-07-0815. PMID 17947483